CLINICAL TRIAL: NCT04636567
Title: A Phase 2 Open-label Study to Evaluate the Use of Nerindocianine as a Surgical Aid in the Delineation of Abdominopelvic Ureter Anatomy Via Near-infrared Fluorescence Imaging in the Setting of Minimally Invasive Surgery
Brief Title: Open-label Study to Evaluate Nerindocianine as a Surgical Aid in Ureter Delineation During Minimally Invasive Surgery
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Clinical program has been suspended for business reasons.
Sponsor: Li-Cor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LICOR-10417-04
Record Dates: First submitted 2020-11-11; First posted 2020-11-19 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2020-11

CONDITIONS: Intraoperative Ureter Injury
Keywords: contrast agent; intraoperative monitoring; intraoperative procedures; near infrared fluorescence; minimally invasive
MeSH Terms: interventions — Injections; IRDye 800BK

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nerindocianine for injection (Experimental): One Arm: Nerindocianine for Injection (0.055 mg/kg body weight); solution, intravenous, one time administration during surgery.
  Interventions: Drug: Nerindocianine for injection

INTERVENTIONS:
Drug: Nerindocianine for injection — Procedure: routine minimally invasive abdominopelvic surgery.
  Other Names: IRDye 800BK

SUMMARY:
Phase 2, multicenter, efficacy and safety study evaluating the use of nerindocianine for the delineation of abdominopelvic ureter anatomy via near infrared fluorescence imaging during minimally invasive lower abdominal surgery (e.g. gynecological, lower gastrointestinal, or other lower abdominal surgery).

DETAILED DESCRIPTION:
The primary objective of this study is to assess the acceptance of near-infrared (NIR) fluorescence imaging (650 to 900 nm) compared to white light (WL) using 3 3-point Likert scales.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent prior to the initiation of study procedures.
* At least 18 years of age.
* Consent to undergo minimally invasive, lower pelvic surgery.

Exclusion Criteria:

* Unwilling or unable to provide informed consent.
* Unwilling or unable to comply with the requirements of the protocol.
* Females who are pregnant, lactating, or planning a pregnancy throughout the study.
* Patients administered indocyanine green (ICG) at the same time of the lower pelvic surgery.
* Have known allergies to D-mannitol and/or citric acid.
* Participation in another clinical trial involving a drug in the past 12 weeks.
* Any other condition that, in the investigator's judgment, would potentially compromise the study compliance or the ability to evaluate safety or efficacy of the investigational product, or determined not a safe candidate for surgery based on standard of care for current medical condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of ureter delineation using a Likert scale to measure ureter visualization | Surgical procedure duration, estimated up to 5 hours
  Evaluation of the pelvic ureter under WL and NIR illumination

SECONDARY OUTCOMES:
Treatment-Emergent Adverse Events | 30 +/- 5 days
  Incidence of Treatment-Emergent Serious Adverse Events and/or Treatment-Emergent Adverse Events
Hourly time point scores concurrence with video review | Scoring occurs at 1-hour intervals for duration of surgical procedure (estimated duration from 1 to 5 hours)
  Three 3-pt Likert scale scores at hourly time points during the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanna Da Silva Southwich, M.D., Principal Investigator — Cleveland Clinic Florida; Jubilee Brown, M.D., Principal Investigator — Carolinas Medical Center / Levine Cancer Institute
Locations (2):
- United States (2):
  - Cleveland Clinic Florida, Weston, Florida
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available.